CLINICAL TRIAL: NCT03048045
Title: Long-term Results After Systematic Periodontal Therapy
Acronym: SYSPERIO10
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Eickholz, Prof. Dr. Peter Eickholz, Goethe University
Other Study IDs: 61/15
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Tooth Loss
Keywords: chronic periodontitis; aggressive periodontitis; supportive periodontal treatment
MeSH Terms: conditions — Tooth Loss; Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supportive Periodontal Treatment (SPT): * at least 18 years old.
  * periodontal treatment (antiinfective therapy with subgingival debridement under local anesthesia and if required periodontal surgery) at the Dept. of Periodontology starting after April 2005 durchgeführt.
  * complete periodontal charting (PPD and PAL-V at 6 sites per tooth, furcation involvement [Hamp et al. 1975] at all furcation sites of multi-rooted teeth) prior to treatment (baseline, T0) and after completion of active periodontal treatment (APT) (reevaluation 1 or 2/start of supportive periodontal therapy, T1)
  * radiographs of all teeth (periapical radiographs or panoramic radiograph) from baseline
  * written informed consent
  Interventions: Procedure: Supportive Periodontal Treatment (SPT)

INTERVENTIONS:
Procedure: Supportive Periodontal Treatment (SPT) — Assessment of Gingival Bleeding Index and Plaque Control Record, re-instruction and re-motivation to effective individual plaque control, professional tooth cleaning, application of a fluoride gel. Twice a year a periodontal charting with probing pocket depths (PPD) and vertical attachment Level (PAL-V) are obtained at 6 sites per tooth. Thirty seconds after probing bleeding on probing (BOP) is recorded. Sites exhibiting PPD = 4 mm and BOP as well as sites with PPD >/= 5 mm are scaled subgingivally. Assignment of SPT intervals is performed according to the periodontal risk assessment (PRA).

SUMMARY:
Patients who had had systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004 are re-examined 10 years +/- 12 months after accomplishment of active periodontal therapy (re-evaluation 1 or 2, start of supportive periodontal treatment) until 100 patients have been enroled. Radiographs (periapicals or panoramics) from start of treatment should be available.

DETAILED DESCRIPTION:
5. Material and Methods

5.1 Patients

Patients who had had systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004 are re-examined 10 years +/- 12 months after accomplishment of active periodontal therapy (re-evaluation 1 or 2, start of supportive periodontal treatment) until 100 patients have been enroled. Radiographs (periapicals or panoramics) from start of treatment should be available.

Inclusion criteria:

* at least 18 years old
* systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia according to the full mouth disinfection protocol and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004
* complete periodontal charts (probing pocket depths [PPD] and vertical probing attachment level [PAL-V] at 6 sites per tooth, furcation involvement at all furcation sites of multi-rooted teeth) Prior to periodontal treatment (baseline, T0) and after accomplishment of active periodontal Treatment (APT) (reevaluation 1 or 2 and start of SPT, T1)
* radiographs of all teeth (periapical or panoramic) at baseline
* written informed consent.

Exclusion citeria:

- Patients that do not meet the inclusion criteria.

Individual dropout criteria:

retraction of consent

5.2 Recruitment and clinical examination

All patients who had had systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia according to the full mouth disinfection protocol and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004 and of whom radiographs (periapicals or panoramics) from start of treatment are available are invited for re-examination 10 years +/- 12 months after accomplishment of active periodontal therapy (re-evaluation 1 or 2, start of supportive periodontal treatment) until 100 patients have been enroled. For patients not agreeing to the invitation the respective reasons are documented (e.g. could not be contacted due to unknown new address). The follow-up is performed by the participating examiners and encompasses the following examinations:

* measurement of CO in exhaled air as measure for cigarette smoking (Bedfont EC50-Micro; Bedfont Scientific Ltd, Rochester, Great Britain). Patients are asked for cigarette smoking: Do you actually smoke and if yes, how many cigarettes per day? Did you smoke in earlier times? If yes how long (years) and how many cigarettes per day? After the questionnaire the CO measurement is repeated.
* Using patients' charts it is documented for each patient whether he or she had attended SPT at the Dept. of Periodontology of the Goethe-University Frankfurt regularly complying with the intervals that had been recommended. If a patient had extended the recommended SPT interval at least once more than 100% he or she is assigned to the irregular SPT group (e.g. the recommended SPT interval is 6 months and the patient returns for SPT after 13 months). Further, rhythm and number of SPT visits is scored.
* General medical history and extended helath questionnaire
* Dental status, sensitivity testing
* Modified GBI
* Modified PCR
* Measurement of probing pocket depths (PPD) and vertical attachment levels (PAL-V) to the nearest 1 mm using a manual periodontal probe (PCPUNC 15; Hu Friedy, Chicago, IL, USA) at 6 sites per tooth, bleeding on probing after 30 s (BOP), and suppuration on probing (SUP). Implantats are measured like teeth but marked as implants.
* At multirooted teeth assessment of furcation involvement using a Nabers probe that was marked in 3 mm increments (PQ2N; Hu Friedy, Chicago, IL, USA)
* Test for interleukin-1 (IL-1) polymorphism (IL-1A -889, IL-1B +3953) (GenoType IL-1-Test, Hain Life Science GmbH, Nehren, Germany), if IL-1 polymorphism had not been tested during routine SPT to estimate the individual periodontal risk and SPT interval. A patient is classified as IL-1 positive if both the second allele for IL-1A and IL-1B are positive.
* All patients who have lost teeth are asked for the reasons (e.g. caries, endodontic, periodontal, orthodontic, prosthetic, trauma etc.).
* All patients were asked about satisfaction with the aesthetic aspects of their periodontal situation (OHIP).

In each patient PPD and PAL-V measurements are repeated in one sextant to assess the reproducibility of measurements.

5.3 Radiographic evaluation

Prior to subgingival debridement/periodontal surgery periapical radiographs (Insight; Kodac, Rochester, NY, USA) using film holders (XCP, Kentzler & Kaschner Dental, Ellwangen/Jagst) or panoramic radiographs had been obtained. Radiographs were obtained using the appropriate dose (Heliodent 70*, 70 kV, 7 mA, Sirona, Bensheim) and were developed (XR24 nova*, Dürr Dental, Bietigheim-Bissingen).

All radiographs are viewed in a darkened room using a radiograph screen. Relative percentage of bone loss is assessed at the most periodontally affected site of each tooth using a Schei ruler. Teeth were assigned i) to one of 5 groups of periodontal bone loss (< 20%, 20/< 40%, 40/< 60%, 60/< 80%, 80% and more) and ii) in conjunction with furcation involvement to one of 3 groups for the assessment of tooth-related prognosis (< 50%, 50-75%, > 75%). Furthermore, at the interproximal site with the most severe bone loss of each tooth, the type of bone loss is characterized as horizontal or vertical (infrabony defect). At each infrabony defect the depth of the infrabony component is measured to the next 0.1 mm using a loupe with 10fold magnification (Scale loupe 10x, Peak, Tohkai Sangyo, Tokyo, Japan). Each infrabony defect is allocated to one of 3 groups: shallow (2 mm), moderate (2.5-4 mm), and deep (>/= 4.5 mm) defects. For each tooth it is assessed whether a double contour of the root could be detected. A double contour is interpreted as indicator for a mesial or distal root groove.

All radiographic assessments are performed by an independent examiner blinded for clinical measurements and therapy rendered.

5.4 Evaluation of patient charts

Each patient is assigned to a periodontal diagnosis (e.g. generalised moderate chronic periodontitis) according to the actual classification of periodontal diseases.

According to baseline data each tooth is assigned to a prognosis category:

* hopeless: bone loss > 75% or the tooth fulfils at least 2 criteria of category "questionable";
* questionable: bone loss between 50 and 75% or infrabony pocket (infrabony component > 2 mm) or furcation involvement;
* good: bone loss < 50% and nonne of the criteria for "qustionable" or "hopeless" are present.

For each patient a prognosis index is calculated (number of hopeless and questionable teeth divided by the whole number of teeth).

The periodontal status at re-examination will be scored according to the most recent criteria of the Swiss Dental Society using precise threshold according to the 2005 criteria.

5.5 Statistical analysis

The patient is defined as statistical unit. Main outcome variable is tooth loss from the end of APT (T1) to re-examination (T2). Secondary endpoints are: PAL-V loss, PISA (periodtally inflamed surface area) change from T1 to T2, SSO criteria at T0, T1, T2 as well as average PPD, PISA, PPD categories at T0, T1, T2.

Using Poisson regression analysis patient-related factors (sex, age, socieconimic status, baseline diagnosis [chronic or aggressive periodontitis], IL-1 polymorphism, mean bone loss in %, cigarette consumption, regular SPT participation ) and using logistic multilevel regression analysis tooth-related (PPD at T1 [deepest pocket/tooth], PAL-V at T1, bone loss in % [T0], furcation involvement [most severe furcation ionvolvement/tooth], tooth type [single-rooted, multi-rooted with/without furcation involvement], type of bone loss [horizontal/vertical, shallow, moderate, deep infrabony defects], baseline prognosis) factors shall be indentified that explain tooth loss during SPT or quality standards.

ELIGIBILITY:
Inclusion criteria:

* at least 18 years old
* systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia according to the full mouth disinfection protocol and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004
* complete periodontal charts (probing pocket depths [PPD] and vertical probing attachment level [PAL-V] at 6 sites per tooth, furcation involvement at all furcation sites of multi-rooted teeth) Prior to periodontal treatment (baseline, T0) and after accomplishment of active periodontal Treatment (APT) (reevaluation 1 or 2 and start of SPT, T1)
* radiographs of all teeth (periapical or panoramic) at baseline
* written informed consent

Exclusion citeria:

* younger than 18 years
* no systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia according to the full mouth disinfection protocol and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004
* missing complete periodontal charts (probing pocket depths [PPD] and vertical probing attachment level [PAL-V] at 6 sites per tooth, furcation involvement at all furcation sites of multi-rooted teeth) Prior to periodontal treatment (baseline, T0) and after accomplishment of active periodontal Treatment (APT) (reevaluation 1 or 2 and start of SPT, T1)
* no radiographs of all teeth (periapical or panoramic) at baseline
* missing written informed consent.

Individual dropout criteria:

- retraction of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had had systematic periodontal treatment (antiinfective treatment with subgingival debridement under local anaesthesia and if required periodontal surgery) at the Dept. of Periodontology starting from October 2004 are re-examined 10 years +/- 12 months after accomplishment of active periodontal therapy (re-evaluation 1 or 2, start of supportive periodontal treatment) until 100 patients have been enroled. Radiographs (periapicals or panoramics) from start of treatment should be available.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
tooth loss during supportive periodontal treatment | 10 years
  tooth loss during supportive periodontal treatment

SECONDARY OUTCOMES:
clinical attachment loss during supportive periodontal treatment | 10 years
  clinical attachment loss during supportive periodontal treatment

OTHER OUTCOMES:
Change of PISA during supportive periodontal treatment | 10 years
  Change of PISA during supportive periodontal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eickholz, Prof. Dr., Study Director — Goethe University
Locations (1):
- Dept. of Periodontology, Center of Dentistry and Oral Medicine, Johann Wolfgang Goethe-University, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petsos H, Ramich T, Nickles K, Dannewitz B, Pfeifer L, Zuhr O, Eickholz P. Tooth loss in periodontally compromised patients: Retrospective long-term results 10 years after active periodontal therapy - tooth-related outcomes. J Periodontol. 2021 Dec;92(12):1761-1775. doi: 10.1002/JPER.21-0056. Epub 2021 May 6. PMID 33748997
- [Result] Petsos H, Schacher B, Ramich T, Nickles K, Dannewitz B, Arendt S, Seidel K, Eickholz P. Retrospectively analysed tooth loss in periodontally compromised patients: Long-term results 10 years after active periodontal therapy-Patient-related outcomes. J Periodontal Res. 2020 Dec;55(6):946-958. doi: 10.1111/jre.12786. Epub 2020 Jul 22. PMID 33145760
- [Result] Graetz C, Baumer A, Eickholz P, Kocher T, Petsos H, Pretzl B, Schwendicke F, Holtfreter B. Long-term tooth retention in periodontitis patients in four German university centres. J Dent. 2020 Mar;94:103307. doi: 10.1016/j.jdent.2020.103307. Epub 2020 Feb 26. PMID 32112911
- [Derived] Schroder M, Buchinger M, Dahmer I, Eickholz P, Petsos H. Clinical Treatment Endpoints After Active Periodontal Treatment and 10 Years of Supportive Periodontal Care: A Retrospective Cohort Study. J Clin Periodontol. 2025 Oct;52(10):1386-1397. doi: 10.1111/jcpe.14179. Epub 2025 Jul 8. PMID 40629762
- [Derived] Vogt L, Pretzl B, Eickholz P, Ramich T, Nickles K, Petsos H. Oral health-related quality of life and patient-reported outcome measures after 10 years of supportive periodontal care. Clin Oral Investig. 2023 Jun;27(6):2851-2864. doi: 10.1007/s00784-023-04876-9. Epub 2023 Feb 1. PMID 36723714